CLINICAL TRIAL: NCT01899326
Title: Pilot Clinical Study of GCSF in Combination With Desipramine for Autologous Stem Cell Mobilization in Multiple Myeloma
Brief Title: Desipramine Hydrochloride and Filgrastim For Stem Cell Mobilization in Patients With Multiple Myeloma Undergoing Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped during the interim analysis due to low accrual after the widespread use of plerixafor for multiple myeloma in the United States.
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amit Verma, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-230; NCI-2013-01212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-010; 2012-230 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: DS (Durie/Salmon) Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Desipramine; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (desipramine, filgrastim) (Experimental): Participants received desipramine hydrochloride PO daily on days -3 to +4 and filgrastim PO BID on days 1-4. Stem cell collection began on day 6.
  Interventions: Drug: Desipramine Hydrochloride; Biological: Filgrastim; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Desipramine Hydrochloride — Given PO
  Other Names: Norpramin; Pertofrane
Biological: Filgrastim — Given PO
  Other Names: G-CSF; Nivestim; r-metHuG-CSF
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studied how well desipramine hydrochloride and filgrastim worked for stem cell mobilization in participants with multiple myeloma (MM) undergoing stem cell transplant. Giving colony-stimulating factors, such as filgrastim, and other drugs, such as desipramine hydrochloride, helps stem cells move from the participant's bone marrow to the blood so they can be collected and stored.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study efficacy, safety, harvest kinetics and engraftment kinetics of participants undergoing autologous stem cell mobilization, mobilized with a combination of granulocyte colony-stimulating factor (GCSF) (filgrastim) with desipramine (desipramine hydrochloride) (G+D).

II. To analyze polymorphisms of adrenergic receptor beta 2 (ADRB2) and adrenergic receptor beta 3 (ADRB3) genes that correlate with mobilization efficiency.

OUTLINE:

Participants received desipramine hydrochloride orally (PO) daily on days -3 to +4 and filgrastim PO twice daily (BID) on days 1-4. Stem cell collection began on day 6.

After completion of study treatment, participants were followed up to 1 week after completion of stem cell collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for autologous stem cell transplant for multiple myeloma; planned use of filgrastim (GCSF) for stem cell mobilization
* Ability to give informed consent
* Glomerular filtration rate (GFR) > 30 ml/minute
* Liver function tests < 2.5 x upper limit of normal (ULN)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2 or less
* Based on prior therapy patients will be classified into two categories:

  * Initial mobilizers with no exposure to alkylators
  * Remobilizers or with prior exposure to alkylators or with greater than 5 cycles of lenalidomide therapy prior to mobilization

Exclusion Criteria:

* Use of a monoamine oxidase inhibitor (MAO-I) during or within 2 weeks of desipramine therapy
* Concomitant therapy with any drugs shown to have major interactions with desipramine
* Concurrent use of drugs that are contraindicated with desipramine
* Myocardial infarction in preceding 4 weeks; history of uncontrolled cardiac arrhythmias or family history of sudden cardiac death; baseline corrected QT (QTc) > 460 msec
* Active alcohol abuse
* Bipolar disorder
* Untreated active major depression
* History of seizures in the past 3 years
* Pregnancy and lactation; refusal to use adequate contraception
* Uncontrolled thyroid disease
* GCSF or pegfilgrastim use within 14 days prior to enrollment
* Bortezomib, Revlimid or thalidomide use within 7 days of enrollment
* Patients with sickle cell disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murali Janakiram, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten participants with multiple myeloma between 18-70 years of age eligible for Autologous Stem Cell Transplant (ASCT) were enrolled in the study between September 2013 and July 2014.
Pre-assignment Details: Of the 10 participants enrolled, 1 participant dropped out after enrollment and prior to study drug initiation. Of the remaining 9 participants, 6 participants underwent stem cell transplantation and completed the full study protocol.
Groups:
- Treatment (Desipramine, Filgrastim): Participants received 100mg desipramine hydrochloride PO daily from Day -3 to Day +4 (8 days total) and filgrastim PO BID from Day +1 to Day +4. Complete blood count (CBC) and peripheral blood CD34+ counts were determined on Day +4 and Day +5. Leukapheresis was started when peripheral blood CD34+ count exceeded 10/uL. If CD34+ counts were <10/uL on Day +5, plerixafor was added as a salvage therapy. Daily leukapheresis was performed with four times the estimated blood volume during each collection until a target cell dose of at least 5x10^6 cells/kg was reached. If the collected CD34+ cell dose was <0.5x10^6 on two consecutive days, aperheris was stopped and the patient was taken off study.
  Despiramine hydrochloride: PO Filgrastim: PO
Period: Overall Study
Arm/Group | Treatment (Desipramine, Filgrastim)
Started | 10
Completed | 6
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Not completed — Disease Relapse (patient with previously undiagnosed relapsing disease) | 1

BASELINE CHARACTERISTICS:
Population: The respective baseline measures were provided for the 6 participants who completed the protocol.
Groups:
- Treatment (Desipramine, Filgrastim): Patients received 100mg desipramine hydrochloride PO daily from Day -3 to Day +4 (8 days total) and filgrastim PO BID from Day +1 to Day +4. Complete blood count (CBC) and peripheral blood CD34+ counts were determined on Day +4 and Day +5. Leukapheresis was started when peripheral blood CD34+ count exceeded 10/uL. If CD34+ counts were <10/uL on Day +5, plerixafor was added as a salvage therapy. Daily leukapheresis was performed with four times the estimated blood volume during each collection until a target cell dose of at least 5x10^6 cells/kg was reached. If the collected CD34+ cell dose was <0.5x10^6 on two consecutive days, aperheris was stopped and the patient was taken off study.
  Despiramine hydrochloride: PO Filgrastim: PO
Arm/Group | Treatment (Desipramine, Filgrastim)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] — Population: Age range of the 6 patients who completed the study.
  years | 59.5 [58 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender of the 6 patients who completed the study.
  Participants
    Female | 4
    Male | 2
Region of Enrollment [Number; unit: participants] — Population: Region of enrollment of the 6 patients who completed the study.
  participants
    United States | 6
Prior Lenalidomide therapy [Count of Participants; unit: Participants] — Number of patients who had received Lenalidomide prior to the trial. Population: Number of patients who had received Lenalidomide prior to the trial who completed the study.
  Participants
    Yes | 4
    No | 2
Prior chemotherapies [Number; unit: participants] — Number of prior chemotherapy treatments. Population: Number of prior chemotherapy treatments for the study participants who completed the trial.
  participants
    One prior chemotherapy treatment | 5
    >1 prior chemotherapy treatment | 1

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Stem Cell Mobilization (SCM) in Participants Who Completed Filgrastim and Desipramine Therapy
Description: Success rate was assessed as the number of participants with Multiple Myeloma (MM) who were first time mobilizers or unexposed to alkylating agents who completed the full course of filgrastim and desipramine and achieved the target collection of >=5 x 10^6 CD34+ cells/kg.
Time Frame: Day 5
Population: 6 participants underwent stem cell transplantation and completed the full study protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Desipramine, Filgrastim): Patients received 100mg desipramine hydrochloride PO daily from Day -3 to Day +4 (8 days total) and filgrastim PO BID from Day +1 to Day +4. Complete blood count (CBC) and peripheral blood CD34+ counts were determined on Day +4 and Day +5. Leukapheresis was started when peripheral blood CD34+ count exceeded 10/uL. If CD34+ counts were <10/uL on Day +5, plerixafor was added as a salvage therapy. Daily leukapheresis was performed with four times the estimated blood volume during each collection until a target cell dose of at least 5x10^6 cells/kg was reached. If the collected CD34+ cell dose was <0.5x10^6 on two consecutive days, apheresis was stopped and the patient was taken off study.
  Despiramine hydrochloride: PO Filgrastim: PO
Arm/Group | Treatment (Desipramine, Filgrastim)
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Success Rate of Stem Cell Mobilization (SCM) in Participants Who Failed Prior Mobilization or Who Were Exposed to Alkylator Therapy or Who Were Predicted to be Difficult to Mobilize Who Completed Filgrastim and Desipramine Therapy
Description: Success rate was assessed as the number of participants with Multiple Myeloma (MM) who Failed Prior Mobilization or who were Exposed to Alkylator Therapy or who were Predicted to be Difficult to Mobilize who completed the full course of filgrastim and desipramine and achieved the target collection of >=5 x 10^6 CD34+ cells/kg.
Time Frame: Day 5
Population: No patients who failed prior mobilization or who were exposed to alkylator therapy or were predicted to be difficult to mobilize were enrolled and as such no data was collected/analyzed for this Outcome Measure.
Arm/Group | Treatment (Desipramine, Filgrastim)
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Number of Days of Apheresis
Description: Median number of days of apheresis required to collect >=5 x 10^6 CD34+ cells/kg. Standard descriptive statistics were used to summarize the data.
Time Frame: Up to 1 week following completion of study treatment, up to 15 days
Population: 6 participants underwent stem cell transplantation and completed the full study protocol.
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Desipramine, Filgrastim)
Number analyzed (Participants) | 6
Days | 1.5 [1 to 2]

4. Secondary Outcome: Incidence of Adverse Events
Description: Incidence of adverse events up to 1 week following completion of study treatment. Adverse events were graded using Version 4.0 of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
Time Frame: Up to 1 week following completion of study treatment, up to 15 days
Population: 6 participants underwent stem cell transplantation and completed the full study protocol.
Measure: Number; unit: Adverse Events
Arm/Group | Treatment (Desipramine, Filgrastim)
Number analyzed (Participants) | 6
Adverse Events | 9

5. Secondary Outcome: Median Time to Neutrophil Engraftment
Description: Median time (number of days) to neutrophil engraftment was determined as first of three consecutive days with absolute neutrophil count (ANC) > 500/ul or first day with ANC > 1000/ul in the absence of growth factor support.
Time Frame: Up to 1 week following completion of study treatment, up to 15 days
Population: 6 participants underwent stem cell transplantation and completed the full study protocol.
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Treatment (Desipramine, Filgrastim)
Number analyzed (Participants) | 6
number of days | 12 [11.8 to 12]

6. Secondary Outcome: Median Time to Platelet Engraftment
Description: Median time (number of days) to platelet engraftment was determined as first of three consecutive days with platelets > 20,000/ul without transfusion.
Time Frame: Up to 1 week following completion of study treatment, up to 15 days
Population: 6 participants underwent stem cell transplantation and completed the full study protocol.
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Treatment (Desipramine, Filgrastim)
Number analyzed (Participants) | 6
number of days | 13.5 [12 to 14.6]

ADVERSE EVENTS:
Time Frame: Subjects were monitored for incidence of Adverse Events up to 1 week following completion of treatment, for a total of up to 15 days
Arm/Group | Treatment (Desipramine, Filgrastim)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Desipramine, Filgrastim) (N=6)
Nausea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Dry Mouth (Skin and subcutaneous tissue disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Target enrollment (n=20) was not reached. The study was stopped during the interim analysis due to low accrual after the widespread use of plerixafor for multiple myeloma in the United States.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes